CLINICAL TRIAL: NCT03377985
Title: Ultrasound Guided Axillary Brachial Plexus Block Versus Supraclavicular Block in Emergency Crushed Hand Patients: A Comparative Study
Brief Title: Ultrasound Guided Axillary Brachial Plexus Block Versus Supraclavicular Block in Emergency Crushed Hand Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: FWA 000017585
Record Dates: First submitted 2017-12-07; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: the Study Focuses on Comparing Between Supraclavicular and Axillary Blocks
MeSH Terms: interventions — Brachial Plexus Block; Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- axillary brachial plexus block group (Active Comparator): Patients placed in the supine position with arm to be blocked abducted and externally rotated. After sterilization of the axilla ultrasound device with high frequency of 8-12 MHZ, linear transducer was put parallel to the anterior axillary fold at axilla to identify the axillary artery, lateral, medial and posterior cords of the brachial plexus in relation to the axillary artery. Lidocaine 1% was infiltrated subcutaneously 1 cm lateral to the probe, 7-10 ml of bupivacaine 0.5% was injected around each cord of the brachial plexus
  Interventions: Procedure: brachial plexus block
- supraclavicular brachial plexus block group (Active Comparator): patients placed in the supine position with the head of the bed elevated 30 degrees and patient's head turned away from the side to be blocked after skin disinfection, ultrasound device was put transversely parallel to and above the middle third of the clavicle, the probe was tilted till identification of the subclavian artery, 1st rib, pleura and brachial plexus lateral to the subclavian artery and above the 1st rib. Lidocaine 1% was infiltrated subcutaneously 1 cm lateral to the lateral side of the probe. A needle was inserted in plane 1 cm lateral to the probe when adjacent to brachial plexus 25 ml of bubivacaine 0.5% was injected around the brachial plexus
  Interventions: Procedure: brachial plexus block

INTERVENTIONS:
Procedure: brachial plexus block
  Other Names: nerve block

SUMMARY:
The current study focused on ultrasound guided brachial plexus block (BPB) which plays an important role in patients with hand trauma either in pain control or for surgical intervention. The brachial plexus can be blocked by several techniques but the most commonly used are the supraclavicular (SCB) and axillary (AXB) blocks. Aim of this study is to compare between the two techniques as regard performance time, needling time, anesthesia related time, block related complications, number of needle pass, and block related pain. 80 patients were allocated randomly into two equal groups, under ultrasound guidance the SCB and AXB were done for the two groups respectively. The needling time, performance time, anesthesia related time, onset time, number of 1st needle pass in each group and block related complications were noted.

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA physical status II and III, and body mass index (BMI) between 20 and 35, aged 40-70, undergoing emergency crushed hand surgery

Exclusion Criteria:

* Patients with significant coagulopathy, infection or trauma at the injection site of local anesthetics, allergy to local anesthetics, refusal to participate, known neuropathies patients, mentally retarded patients, severely trauma patients who required general anesthesia from the start in the pre-induction room, and unconscious patients due to the accident. Also, shocked patients and patients with chronic obstructive airway disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
block related complications | 24 hours after the block
  failed block, motor weakness 24 h after the block, vascular puncture, Horner syndrome, paresthesia and pneumothorax

SECONDARY OUTCOMES:
number of first needle pass | 10-20 min
  how many times the needle is inserted till we can inject local anesthesia in a proper site